CLINICAL TRIAL: NCT06762093
Title: Management and Outcomes of Traumatic Eyelid Injuries in Assiut University Hospital
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Ismail Moussa Abdellateef, Residant doctor at Assiut university hospital, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Traumatic Eyelid Injuries MO
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Traumatic Eyelid Injuries
MeSH Terms: interventions — Wound Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- traumatic eyelid injuries (Active Comparator): * Patients of all ages presenting with traumatic eyelid injuries to the study institution in either ophthalmology or emergency departments.
  * Traumatic eyelid injuries can include, but are not limited to:
    * Contusions
    * Lacerations
    * Avulsions
    * Eyelid margin defects
    * Eyelid margin involvement
    * Eyelid crease disruption
    * Eyelid tissue loss
  Interventions: Procedure: surgical repaire

INTERVENTIONS:
Procedure: surgical repaire — * Primary closure of lacerations
  * Eyelid margin repair
  * Eyelid crease reconstruction
  * Eyelid transposition flaps or grafts
  * Tarsorrhaphy
  Other Names: Surgical Repair

SUMMARY:
this study aim To determine the incidence of traumatic eyelid injuries presenting to a tertiary eye care center.

To describe the clinical characteristics of traumatic eyelid injuries, including the etiology, location, and extent of injury.

To evaluate the management approaches utilized for traumatic eyelid injuries, including surgical repair, medical therapy, and other treatments.

To assess the outcomes of traumatic eyelid injuries, including functional outcomes, cosmetic results, and complication rates

DETAILED DESCRIPTION:
Vision is the most cared-for function of the human body, and the eyelids are provided to cover the eye for protection. Eyelids are not only protective curtains in front of the eyes but also contribute to the shape and beauty of the face. They are complex structures designed to protect the globe from various external trauma . Eyelids help to keep the corneas moist, protect against injury and excessive light, and regulate the amount of light reaching the retina. They are essential for the distribution and drainage of tears .

Traumatic eyelid injuries are a common occurrence and can range in severity from minor lacerations to more complex injuries involving the eyelid structures. These injuries can significantly impact a patient's visual function and cosmetic appearance. Understanding the epidemiology, clinical presentation, management approaches, and outcomes of traumatic eyelid injuries is important for optimizing patient care.

Eyelid injuries are an important subtype of facial trauma, which necessitates the ophthalmologist being competent and fully informed . Lacerated wounds of the eyelids are common features of ocular trauma and often occur in isolation without any associated intraocular injuries . Eyelid lacerations can be treated using different techniques depending on their depth, width, injury mechanism, and accompanying injuries. They can be repaired with primary closure, skin flap, or skin graft. Small defects limited to the skin of the eyelids can be repaired by direct closure .

Eyelid trauma may often appear trivial but can have profound effects on injury-associated morbidity. Recovery of full eyelid function and maintenance of the lacrimal apparatus are important considerations when approaching lid trauma [. Proper information and education can help individuals to avoid eye injuries and their substantial burden .

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages presenting with traumatic eyelid injuries to the study institution in either ophthalmology or emergency departments

Exclusion Criteria:

* Patients presented with eyelid injuries who are:
* Presented late
* Presented after a previous intervention
* Known to have co-existing eyelid pathology (as tumors, infections, congenital abnormalities)
* Patients with incomplete medical records or loss to follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
incidence of traumatic eyelid injuries | 2 year
  To determine the incidence of traumatic eyelid injuries presenting to a tertiary eye care center.

IPD SHARING:
Plan to Share IPD: Undecided